CLINICAL TRIAL: NCT04859751
Title: An Open-Label, Single Arm, Multicenter Study to Evaluate the Efficacy and Safety of Intravesical VB4-845 Injection in Patients With Non-Muscle Invasive Bladder Cancer
Brief Title: Study of VB4-845 Injection for Treating Patients With Non-muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB4-845-CN-001
Record Dates: First submitted 2021-04-13; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Non-Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — VB4-845

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VB4-845 Injection (Experimental): Induction - 30 mg of Vicinium in 50 mL of saline administered twice weekly (BIW) for 6 weeks followed by once weekly for 6 weeks, for a total of 12 weeks.
  Maintenance - 30 mg of Vicinium in 50 mL of saline administered once weekly every other week for up to 104 weeks.
  Interventions: Drug: VB4-845 Injection

INTERVENTIONS:
Drug: VB4-845 Injection — Intravesical administration of VB4-845 Injection.

SUMMARY:
Because of the high risk for development of muscle invasive disease, cystectomy is recommended for CIS, high-grade Ta and T1 patients who experience disease recurrence following intravesical therapy. VB4-845 injection is an experimental agent that may provide an alternative to cystectomy

DETAILED DESCRIPTION:
Bladder cancer is the 6th most common cancer in the United States, affecting more men than women. The usual first treatment for NMIBC (Ta, T1,and CIS) is transurethral resection of the bladder tumors followed by intravesical immunotherapy, most commonly with bacillus Calmette-Guérin (BCG).

Because of the high risk for development of muscle invasive disease, cystectomy is recommended for CIS and high-grade Ta and T1 patients who experience disease recurrence following intravesical therapy. For patients unable or unwilling to undergo cystectomy, treatment options are limited.

VB4-845 injection is a recombinant fusion protein produced in Escherichia coli (E. coli) that expresses a humanized single-chain antibody fragment specific for the epithelial cell adhesion molecule (EpCAM) antigen linked to exotoxin A (ETA[252-608]). Once bound to the EpCAM antigen on the surface of carcinoma cells, Vicinium is internalized through an endocytic pathway. The ETA(252-608) is cleaved off and induces cell death by irreversibly blocking protein synthesis.

This is an open-label, non-randomized, multicenter bridging study in Chinese patients with NMIBC, specifically CIS (with or without papillary disease), high-grade Ta or any grade T1 papillary disease, who have previously failed BCG treatment (i.e., not those who are intolerant) with or without interferon. The study consists of a Screening period, a 12-week Induction Phase, and a Maintenance Phase of up to 21 monthly cycles for a total treatment period of up to104 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed non muscle-invasive urothelial carcinoma (transitional cell carcinoma) of the bladder.
2. Subjects must have received adequate BCG treatment defined as at least 2 courses of BCG, i.e., at least one induction and one maintenance course or at least 2 induction courses.
3. The subject's disease is refractory or has relapsed following adequate BCG treatment.
4. Male or non-pregnant, non-breastfeeding female, age 18 years or older at date of consent.
5. All women of childbearing potential (WOCBP) must have a negative pregnancy test within 7 days of the first dose of study therapy.
6. All sexually active subjects agree to use barrier contraception (i.e., condoms) while receiving study treatment and for 120 days following their last dose of study treatment.
7. Karnofsky performance status ≥ 60.
8. Ability to understand and sign an Independent Ethics Committee-or Institutional Review Board-approved informed consent document.

Exclusion Criteria:

1. The subject is pregnant or breastfeeding.
2. Evidence of urethral or upper tract transitional cell carcinoma (TCC) within the past 2 years.
3. Subjects with hydronephrosis, except for those subjects where hydronephrosis has been longstanding and diagnostic evaluation at Screening shows no evidence of tumor.
4. Any intravesicular or other chemotherapy treatment within 2 weeks or any investigational agent within 4 weeks prior to the initial dose of study drug.
5. History of recurrent severe urinary tract infections (UTIs) per investigator judgment. Subjects with a current UTI requiring antibiotic treatment may defer the initiation of Vicinium treatment on Day 1 until resolution of the UTI.
6. he subject has a diagnosis of another malignancy within 2 years before the first dose of study treatment.
7. A QTc interval of >470 msec by the Fridericia formula (QTcF), at the Screening ECG.
8. Subjects who, in the opinion of the Investigator, cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy, biopsy) due to the presence of serious comorbid condition(s).
9. Local or severe allergy to any components of the drug regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | up to 6 months
  Complete response rate in patients with CIS with or without resected papillary disease following initiation of VB4-845 injection therapy

SECONDARY OUTCOMES:
Recurrence-free rate | up to 6 months
  Recurrence-free (RF) rate in patients with high-grade Ta or any grade T1 papillary disease (without CIS)
Complete response rate | up to 3 months
  Complete response rate in patients with CIS with or without resected papillary disease following initiation of VB4-845 injection therapy
Recurrence-free rate | up to 3 months
  Recurrence-free (RF) rate in patients with high-grade Ta or any grade T1 papillary disease (without CIS)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Every 4 weeks up to 104 weeks
  Frequency and severity of adverse events. Including adverse events (AEs), change in physical examination findings, change in vital signs, clinical laboratory testing for systemic safety,including liver function, renal function, compelete blood count, and clinical chemistries.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, PI, Principal Investigator — Shanghai Fudan University Affiliated Tumor Hospital
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No